CLINICAL TRIAL: NCT06018597
Title: The Relationship of Sevoflurane Consumption With Metabolic Age
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, DUYGU DEMİROZ, associate professor, Inonu University
Other Study IDs: Inonu 2022/92
Record Dates: First submitted 2023-08-09; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Sevoflurane
Keywords: Sevoflurane Consumption, Metabolic Age, Tanita
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- percent age difference < -6.6%: The percentage age difference in the negative direction represents patients whose metabolic age is greater than their chronological age.
  When we analyze the ROC analysis in the negative direction,between Percent Age Difference and Sevoflurane Consumption Amount Calculated According to Metabolic Age, the cut-off value of the percentage age difference is -6,6%.
  This group refers to those whose percentage age difference is less than -6.6%
  Interventions: Drug: Sevoflurane Baxter, 100%, Inhalation Vapour, Liquid 250 mL
- percent age difference -6.6% to 11.7% those between: When we analyze the ROC analysis in the negative direction,between Percent Age Difference and Sevoflurane Consumption Amount Calculated According to Metabolic Age, the cut-off value of the percentage age difference is -6,6%. When we analyze the ROC analysis in the positive direction, the cut-off value of the percent age difference is 11.7%.
  This group refers to those whose percentage age difference between -6.6% and 11.7%
  Interventions: Drug: Sevoflurane Baxter, 100%, Inhalation Vapour, Liquid 250 mL
- percent age difference > 11.7%: the percent age difference in the positive direction represents patients whose metabolic age is less than their chronological age.
  When we analyze the ROC analysis in the positive direction,between Percent Age Difference and Sevoflurane Consumption Amount Calculated According to Metabolic Age, the cut-off value of the percent age difference is 11.7%.
  This group refers to those whose percentage age difference is more than 11.7%
  Interventions: Drug: Sevoflurane Baxter, 100%, Inhalation Vapour, Liquid 250 mL

INTERVENTIONS:
Drug: Sevoflurane Baxter, 100%, Inhalation Vapour, Liquid 250 mL — No procedure was performed on the patient other than routine anesthesia management.We compared sevoflurane consumption amount in the patient undergoing general anesthesia with sevoflurane according to their metabolic age.
  Other Names: No procedure was performed on the patient other than routine anesthesia management.

SUMMARY:
The aim of this clinical study is to determine the consumption of sevoflurane, which is one of the inhalation anesthetics, with metabolic age and basal metabolic rate. The basal metabolic rates and metabolic ages of the patients who will be given sevoflurane- maintained general anesthesia were measured preoperatively. The relationship between the amount of sevoflurane consumption and the measured data of the patients in the postoperative period was examined.

DETAILED DESCRIPTION:
Standard monitoring, BIS, TOF (train of four) were performed from the premedication application. Aspect A 2000 (Aspect Medical Systems, Newton) monitor and single-chip BIS electrodes will be used for BIS. The total amount of sevoflurane consumed and MAK values of these components will be recorded. Chronological age, metabolic age, BMR, height, weight, ideal body weight, BMI, body adiposity, body fluid ratio, body fluid care, fat mass, lean body weight, muscle registered, visceral adiposity, obesity degree in the preoperative period of the patients. Values, ASA scores and demographic data will be recorded for the operation process, cutting time, anesthesia time, extubation time, total sevoflurane consumption throughout the case, and the relationship with basal metabolism and metabolic age will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 18-65 who are scheduled for rhinoplasty or septoplasty with ASA I-II Cases lasting 1 to 3 hours

Exclude Criteria:

Patients at high risk of malignant hyperthermia, with a history of allergy to general anesthesia or any of the drugs to be used in the study, accepted as ASA III- ASA IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ALL CENDER
Study Population: 18-65 AGE
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
consumption of sevoflurane | patients during surgery
  Reducing patients' consumption of sevoflurane according to metabolic law

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu universitesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St-Onge MP, Gallagher D. Body composition changes with aging: the cause or the result of alterations in metabolic rate and macronutrient oxidation? Nutrition. 2010 Feb;26(2):152-5. doi: 10.1016/j.nut.2009.07.004. Epub 2009 Dec 8. PMID 20004080
- [Background] Ng JCM, Schooling CM. Effect of Basal Metabolic Rate on Cancer: A Mendelian Randomization Study. Front Genet. 2021 Sep 9;12:735541. doi: 10.3389/fgene.2021.735541. eCollection 2021. PMID 34567085